CLINICAL TRIAL: NCT00205114
Title: Dane County Safety Assessment for Elders (SAFE) Research Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 2003-042
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2007-12

CONDITIONS: Falls

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Individualized multifactorial intervention for community-living high-risk older adults
Behavioral: Health professional education program about fall prevention

SUMMARY:
This 3-year collaborative project will develop, implement, and test a comprehensive approach to the prevention of falls among high-risk older adults in Dane County, Wisconsin through two complementary strategies:

1. a targeted strategy of an individualized multifactorial intervention for community-living high-risk older adults. Older adults are defined as aged 65 and older. High risk is defined as two or more falls in the year prior, one fall with injury, or one fall with gait and balance problems, as per recent guidelines from the American Geriatric Society (AGS). The multifactorial intervention consists of an in-home assessment followed by recommendations to the participant and his/her physician, a prescription for physical therapy, other referrals (optometry, podiatry, occupational therapy, etc.) based on the assessment, monthly phone follow-up for 11 months, and a prescription for long-term exercise after physical therapy.
2. a program to educate primary care physicians, physician assistants, nurse practitioners, and physical therapists in Dane County in the current diagnosis and treatment recommendations for fall prevention.

DETAILED DESCRIPTION:
The purposes of the project are:

1. To test, in a randomized, controlled, single-blind study design, whether a multifactorial intervention for high-risk older adults will decrease the rate of falls compared to a control group receiving a home safety and nutrition booklet by mail;
2. To enhance existing health professional knowledge base to support fall prevention;
3. To test, in a quasi-experimental study design, the ability of a community-wide health professional educational program to decrease the rate of fall-related hospitalizations among older adults (both high and low-risk) in Dane County compared to control counties in Wisconsin.

We hypothesize that:

The rate of falls will be 40% lower over one year among high-risk older adults randomized to the individualized multifactorial intervention (combined with health professional education), compared to those randomized to home safety and nutrition booklets (combined with health professional education) in Dane County.

A health professional education program about fall prevention will decrease the rate of fall-related hospitalizations among older adults (both high and low-risk) in the intervention county by 10%, compared to an anticipated no change from baseline in control counties.

ELIGIBILITY:
Inclusion Criteria:

* Community-residing in Dane County or surrounding communities.
* Seniors living in assisted-living senior apartments
* Aged 65 and older
* At high risk for falls as defined by AGS criteria (two or more falls in the past year, or one fall with injury, or one fall with abnormal gait or balance)

Exclusion Criteria:

* Reside in a community-based residential facility (i.e. group home)
* Are unable to give informed consent and have no related, in-home caregiver

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 500 (Actual)
Dates: Start 2003-12; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Rate of falls among high-risk older adults randomized to the individualized multifactorial intervention | over one year

SECONDARY OUTCOMES:
Rate of fall-related hospitalizations among older adults in the intervention | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Mahoney, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States